CLINICAL TRIAL: NCT03915548
Title: A Phase III, Randomized, Single Blind, Attention Controlled, Multi-center Study of the Effects of a Rehabilitation Intervention on Participation Restrictions of Female Breast Cancer Survivors
Brief Title: Optimizing Functional Recovery of Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen Lyons, ScD, OTR/L, Professor, MGH Institute of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021P002871; 1R01CA225792-01A1 (NIH)
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: The investigators will recruit 300 women over the age of 18 reporting participation restrictions after completing curative treatment for Stage 1-3 breast cancer within the past year. Half of the participants will be randomized to the 4-month BA/PS intervention which consists of 6 weekly telephone calls followed by 3 monthly telephone calls. BA/PS is designed to teach problem-solving and action planning to promote functional recovery. The other half of participants will be assigned to an attention control condition providing education about survivorship topics. This control condition will allow us to account for the effect of time and history, and the non-specific effects of attention
Who Masked: Outcomes Assessor
Masking Description: Assessments will be administered via telephone by a research assistant blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Behavioral Activation/ Problem Solving Intervention (Experimental): BA/PS teaches survivors to a) systematically examine the reasons an activity is challenging, b) set achievable short-term goals that have the potential to improve participation, c) brainstorm solutions including activity adaptations and environmental modifications, d) construct and implement a detailed action plan, and e) evaluate the results and level of goal attainment. The structured process gives participants repeated practice in goal reengagement that leads them progressively closer to their long-term functional goals. The BA/PS framework integrates the cognitive-behavioral therapies of Behavioral Activation and Problem-solving Treatment and incorporates concepts from an occupational therapy theory called the Person-Environment-Occupational Performance Model.
  Interventions: Behavioral: The Behavioral Activation/ Problem Solving Intervention
- Attention Control Condition (Active Comparator): Investigators provide education regarding nine cancer survivorship topics (i.e., healthy diets, physical activity, lymphedema management, smoking cessation, stress management, communication with providers, body image and sexuality, communication with social supports, work accommodations) during the control telephone contacts. The control condition will match the intervention in terms of the number of sessions, the delivery by telephone, use of an occupational therapist, and the use of "homework" between sessions (i.e., reading the education materials for the control condition versus executing the action plan for the BA/PS condition).
  Interventions: Behavioral: Attention Control Condition

INTERVENTIONS:
Behavioral: The Behavioral Activation/ Problem Solving Intervention — The interventionist presents the rationale for BA/PS, promotes a positive problem orientation, and educates about the framework for problem-solving and action planning. The interventionist then administers the Canadian Occupational Performance Measure to elicit participant priorities, motivation, and long-term goals. The interventionist then guides the participant in using the BA/PS framework to set a goal, brainstorm solutions to challenges, and create a detailed action plan for the coming week.
  Arms: The Behavioral Activation/ Problem Solving Intervention
Behavioral: Attention Control Condition — The interventionist provides education regarding nine cancer survivorship topics (i.e., healthy diets, physical activity, lymphedema management, smoking cessation, stress management, communication with providers, body image and sexuality, communication with social supports, work accommodations) during the control telephone contacts.
  Arms: Attention Control Condition

SUMMARY:
This study is a randomized controlled trial (RCT) to test the efficacy of a Behavioral Activation and Problem Solving (BA/PS) approach to improving activity participation over time as compared to an attention control condition within a sample of 300 breast cancer survivors reporting reduced activity participation after completing cancer treatment.

DETAILED DESCRIPTION:
Assessments will be administered via telephone by a research assistant blind to group assignment. Participants will complete outcome assessments upon enrollment (T1) and at 8 weeks (T2), 20 weeks (T3) and 44 weeks (T4) later. The T2 assessment captures the short-term outcomes of the most intensive part of the intervention (i.e., after six weekly sessions). The T3 assessment will capture the short-term outcomes at the end of the full intervention. The T4 assessment explores the sustained effect of BA/PS (six months after BA/PS ends). The study aim is to test whether the BA/PS intervention affects the "slope" of functional recovery over time. With the longitudinal data, the investigators will also be able to explore the pace of improvement and whether the two groups differ at these clinically relevant time points.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older.
2. Experiencing reduced participation (i.e., a score greater than or equal to 10 on the Work and Social Adjustment Scale).
3. Females diagnosed with Stage 1-3 breast cancer and within one year of completion of locoregional treatment and/or chemotherapy with curative intent and absence of disease recurrence

Exclusion Criteria:

1. Non-English speaking.
2. Non-correctable hearing loss.
3. Moderate-severe cognitive impairment indicated by a score < 3 on a 6-item cognitive screener.
4. History of severe mental illness (i.e., schizophrenia, bipolar disorder), current major depressive disorder, active suicidal ideation, or active substance misuse documented within the medical record.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Lyons, ScD, Principal Investigator — MGH Institute of Health Professionals
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyons KD, Wechsler SB, Ejem DB, Stevens CJ, Azuero A, Khalidi S, Hegel MT, Dos Anjos SM, Codini ME, Chamberlin MD, Morency JL, Coffee-Dunning J, Thorp KE, Cloyd DZ, Goedeken S, Newman R, Muse C, Rocque G, Keene K, Pisu M, Echols J, Bakitas MA. Telephone-Based Rehabilitation Intervention to Optimize Activity Participation After Breast Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e242478. doi: 10.1001/jamanetworkopen.2024.2478. PMID 38517442
- [Derived] Stevens CJ, Hegel MT, Bakitas MA, Bruce M, Azuero A, Pisu M, Chamberlin M, Keene K, Rocque G, Ellis D, Gilbert T, Morency JL, Newman RM, Codini ME, Thorp KE, Dos Anjos SM, Cloyd DZ, Echols J, Milford AN, Ingram SA, Davis J, Lyons KD. Study protocol for a multisite randomised controlled trial of a rehabilitation intervention to reduce participation restrictions among female breast cancer survivors. BMJ Open. 2020 Feb 13;10(2):e036864. doi: 10.1136/bmjopen-2020-036864. PMID 32060166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between August 2019 and April 2022. Participants were recruited via Dartmouth College, the University of Alabama at Birmingham (UAB), and via Facebook.
Pre-assignment Details: 19 participants were enrolled and then excluded from the study before assignment to groups. 2 were excluded due to screen failure and 17 were excluded because they did not complete the baseline assessment.
Period: Overall Study
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Started | 144 | 140
Session 1 | 139 | 136
Session 2 | 138 | 135
Session 3 | 134 | 132
Session 4 | 131 | 130
Session 5 | 128 | 128
Session 6 | 127 | 126
Follow-up Data Collection 1 (Week 8) | 124 (8 participants missed data collection time point 12 participants withdrew) | 128 (7 participants missed data collection time point 5 participants withdrew)
Session 7 | 126 | 124
Session 8 | 126 | 119
Session 9 | 120 | 119
Follow-up Data Collection 2 (Week 20) | 123 (4 participants missed data collection time point 5 participants withdrew) | 124 (6 participants missed data collection time point 5 participants withdrew)
Follow-up Data Collection 3 (Week 44) | 118 (9 participants withdrew) | 113 (17 participants withdrew)
Completed (All 144 intervention participants and all 140 control participants were included in the final analyses) | 118 | 113
Not Completed | 26 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition | Total
Number analyzed (Participants) | 144 | 140 | 284
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (9.9) | 56.2 (10.6) | 56.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 140 | 284
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 140 | 138 | 278
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 29 | 47
  White | 124 | 110 | 234
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 144 | 140 | 284
Employment Status [Count of Participants; unit: Participants]
  Employed (FT/PT) | 75 | 77 | 152
  Homemaker/Retired | 42 | 35 | 77
  On Short/Long Term Disability | 12 | 13 | 25
  Unemployed | 10 | 12 | 22
  Other | 3 | 3 | 6
  Missing | 2 | 0 | 2
Education Level [Count of Participants; unit: Participants]
  Some High school/High school Graduate | 9 | 18 | 27
  Some College (2 year) | 35 | 30 | 65
  Graduate (4 year, Master's, Doctoral) | 98 | 92 | 190
  Missing | 2 | 0 | 2
Marital Status [Count of Participants; unit: Participants]
  Never Married | 8 | 11 | 19
  Married/Living with a partner | 98 | 89 | 187
  Separated/Divorced | 32 | 33 | 65
  Widowed | 5 | 7 | 12
  Missing | 1 | 0 | 1
Number of Dependent Children Living at Home [Count of Participants; unit: Participants]
  0 | 103 | 95 | 198
  1 | 21 | 21 | 42
  2 | 15 | 16 | 31
  3 | 3 | 6 | 9
  4 | 1 | 2 | 3
  Missing | 1 | 0 | 1
Insurance Status [Count of Participants; unit: Participants]
  Other/None, Self pay | 4 | 8 | 12
  Medicaid/Medicare, or other government insurance | 37 | 41 | 78
  Private through employer | 96 | 85 | 181
  Missing | 7 | 6 | 13
Household Income [Count of Participants; unit: Participants]
  Less than $40,000 per year | 28 | 32 | 60
  $40,000 per year or more | 114 | 106 | 220
  Missing | 2 | 2 | 4
Rurality [Count of Participants; unit: Participants]
  Urban | 95 | 86 | 181
  Rural | 44 | 49 | 93
  Missing | 5 | 5 | 10
Cancer Stage [Count of Participants; unit: Participants] — Cancer stage was self-reported by participants who were recruited via Facebook, and for all other participants, it was collected via electronic medical record review. Higher stage indicates more advanced disease state.
  Participants
    Stage I | 55 | 64 | 119
    Stage II | 60 | 53 | 113
    Stage III | 29 | 23 | 52
Cancer Treatment [Count of Participants; unit: Participants]
  Surgery | 143 | 139 | 282
  Radiation | 118 | 100 | 218
  Chemotherapy | 96 | 90 | 186
Time Since End of Primary Cancer Treatment [Count of Participants; unit: Participants]
  <6 months | 82 | 81 | 163
  >6 months | 62 | 59 | 121
Disability Days [Mean (Standard Deviation); unit: Days]
  Days Miss Work | 3 (6) | 2.1 (4.5) | 2.5 (5.3)
  Days in Bed | 2.8 (5.3) | 4.2 (7.3) | 3.5 (6.4)
PROMIS: Satisfaction with Social Roles & Activities [Mean (Standard Deviation); unit: T-score] — The Patient Reported Outcomes Measurement Information System (PROMIS): Satisfaction with Social Roles and Activities measures satisfaction with daily routines and activities. Raw scores were converted to T-scores (mean = 50, SD = 10) with higher scores indicating better outcomes (i.e., greater satisfaction with daily routines and activities).
  T-score | 45.6 (6.5) | 45.8 (6.9) | 45.7 (6.7)
PROMIS: Ability to Participate in Social Roles & Activities [Mean (Standard Deviation); unit: T-score] — The Patient Reported Outcomes Measurement Information System (PROMIS): Ability to Participate in Social Roles and Activities measures self-reported ability to participate in daily routines and activities. Raw scores were converted to T-scores (mean = 50, SD = 10) with higher scores indicating better outcomes (i.e., greater ability to participate in daily routines and activities).
  T-score | 43.4 (5.2) | 43.3 (5.5) | 43.3 (5.3)
Work Limitations Questionnaire scale score [Mean (Standard Deviation); unit: units on a scale] | 34.5 (17.4) | 36.0 (19.3) | 35.3 (18.3)
Quality of Life, FACT-G [Mean (Standard Deviation); unit: units on a scale] — The Functional Assessment of Cancer Treatment (FACT) - General measures quality of life. The physical, social, and functional subscale scores can range 0-28 and the emotional subscale score can range 0-24; higher scores indicate better well-being. Overall score was calculated by summing the four subscales; overall scores can range from 0-108 with higher scores indicating better quality of life.
  units on a scale
    Physical | 17 (5.5) | 17 (5.2) | 17.0 (5.3)
    Social | 19.9 (5.2) | 19.1 (6.5) | 19.5 (5.9)
    Emotional | 15.9 (4.5) | 15.8 (4.6) | 15.9 (4.6)
    Functional | 16.5 (5.3) | 16.2 (5.3) | 16.4 (5.3)
    Overall Score | 69.3 (16.3) | 68.1 (17.5) | 68.7 (16.9)
Brief COPE [Mean (Standard Deviation); unit: units on a scale] — Range for each subscale (positive reframing, active coping, planning): 2-8; higher values indicate more adaptive coping. Subscales items are summed; no total score.
  units on a scale
    Active coping | 6.3 (1.5) | 6.5 (1.6) | 6.4 (1.6)
    Planning | 6.3 (1.7) | 6.6 (1.6) | 6.4 (1.7)
    Positive reframing | 6.4 (1.7) | 6.6 (1.7) | 6.4 (1.7)
Goal Adjustment Scale [Mean (Standard Deviation); unit: units on a scale] — Scores range from 4-20 for the goal disengagement subscale and 6-30 for goal reengagement subscale; higher scores indicate greater tendency to disengage or re-engage with goals.
  units on a scale
    Disengagement | 10 (2.9) | 10.9 (3.3) | 10.4 (3.1)
    Reengagement | 21.5 (3.8) | 21.2 (3.9) | 21.3 (3.9)
Hospital Anxiety Depression Scale (HADS) [Mean (Standard Deviation); unit: units on a scale]
  Anxiety | 9.4 (4.3) | 9.0 (4.3) | 9.2 (4.3)
  Depression | 6.0 (3.5) | 6.7 (4.1) | 6.3 (3.8)
Work and Social Adjustment Scale (WASA) score [Mean (Standard Deviation); unit: units on a scale] — The Work and Social Adjustment Scale (WASA) measures self-reported disability; higher score indicating greater disability. Scores range 0-40.
  units on a scale | 16.3 (6.5) | 17.5 (7.1) | 16.9 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Participation Satisfaction in Social Roles and Activities: PROMIS
Description: The Patient Reported Outcomes Measurement Information System (PROMIS): Satisfaction with Social Roles and Activities measures satisfaction with daily routines and activities. Raw scores (ranging 8-40) were converted to T-scores (mean = 50, SD = 10) with higher scores indicating better outcomes (i.e., greater satisfaction with daily routines and activities).
Time Frame: The overall treatment effect will be computed as the between-group differences at weeks 8, 20, 44 (adjusted for baseline) estimated with a linear contrast.
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
T-score
  Week 0 | 45.75 (.43) | 46 (.44)
  Week 8: number analyzed (Participants) | 124 | 128
  Week 8 | 48.09 (.47) | 47.61 (.46)
  Week 20: number analyzed (Participants) | 123 | 124
  Week 20 | 50.47 (.47) | 49.81 (.47)
  Week 44: number analyzed (Participants) | 118 | 113
  Week 44 | 50.85 (.48) | 51.39 (.49)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = .54, Mixed Models Analysis — Adjusted; multiple-degree-of-freedom test; F(3,747)=0.88

2. Primary Outcome: Participation Ability in Social Roles and Activities
Description: The Patient Reported Outcomes Measurement Information System (PROMIS): Ability to Participate in Social Roles and Activities Short Form 8a measures participation with daily routines and activities. Raw scores (ranging 8-40) were converted to T-scores (mean = 50, SD = 10) with higher scores indicating better outcomes (i.e., greater ability to participate in daily routines and activities).
Time Frame: The overall treatment effect will be computed as between-group differences at weeks 8, 20, 44 (adjusted for baseline), estimated with a linear contrast.
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: T-scores
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
T-scores
  Week 0 | 43.55 (.4) | 43.48 (.41)
  Week 8: number analyzed (Participants) | 124 | 128
  Week 8 | 45.55 (.43) | 44.95 (.43)
  Week 20: number analyzed (Participants) | 123 | 124
  Week 20 | 47.27 (.43) | 46.44 (.43)
  Week 44: number analyzed (Participants) | 118 | 113
  Week 44 | 47.43 (.44) | 48.63 (.45)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = .09, Mixed Models Analysis — Adjusted; multiple-degree-of-freedom test; F(3,746.4)=2.64

3. Primary Outcome: Productivity
Description: Instrument name: Disability Days section of the Medical Expenditure Panel Survey (MEPS).
  Range: 0- 30 days. Subscales: N/A. Interpretation: Higher values indicate lower productivity.
Time Frame: as for outcome 1
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: days
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
days
  Week 0 | 1.32 (.17) | 1.15 (.15)
  Week 8: number analyzed (Participants) | 124 | 128
  Week 8 | 1.03 (.14) | .91 (.12)
  Week 20: number analyzed (Participants) | 123 | 124
  Week 20 | 1.22 (.16) | .87 (.12)
  Week 44: number analyzed (Participants) | 118 | 113
  Week 44 | .88 (.13) | .76 (.11)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = .55, Mixed Models Analysis — Adjusted; Poisson model with log link; multiple-degree-of-freedom test; F(3,717)=0.7

4. Primary Outcome: Work Productivity
Description: The Work Limitations Questionnaire-Short Form (WLQ-SF) assesses productivity with an overall score indicating the percentage decrement in productivity in the previous two weeks. Scores range 0-100% with higher scores indicating greater decrement in productivity.
Time Frame: The overall treatment effect will be computed as the between-group differences at weeks 8, 20, 44 (adjusted for baseline), estimated with a linear contrast.
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
score on a scale
  Week 0 | 34.7 (1.58) | 34.15 (1.6)
  Week 8: number analyzed (Participants) | 124 | 128
  Week 8 | 27.87 (1.71) | 25.35 (1.67)
  Week 20: number analyzed (Participants) | 123 | 124
  Week 20 | 25.13 (1.73) | 23.57 (1.69)
  Week 44: number analyzed (Participants) | 118 | 113
  Week 44 | 22.79 (1.73) | 21.14 (1.75)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = .99, Mixed Models Analysis — Adjusted; multiple-degree-of-freedom test; F(3,394.7)=0.18

5. Secondary Outcome: Quality of Life: Functional Assessment of Cancer Therapy- (FACT-G)
Description: The Functional Assessment of Cancer Treatment (FACT) - General measures quality of life. The physical, social, and functional subscale scores can range 0-28 and the emotional subscale score can range 0-24; higher scores indicate better well-being. Overall score was calculated by summing the four subscales; overall scores can range from 0-108 with higher scores indicating better quality of life.
Time Frame: as for outcome 4
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
score on a scale
  Overall score: Week 0 | 69.66 (.87) | 69.45 (.89)
  Overall score: Week 8: number analyzed (Participants) | 124 | 128
  Overall score: Week 8 | 73.44 (.93) | 73.36 (.92)
  Overall score: Week 20: number analyzed (Participants) | 123 | 124
  Overall score: Week 20 | 76.25 (.93) | 76.49 (.93)
  Overall score: Week 44: number analyzed (Participants) | 118 | 113
  Overall score: Week 44 | 76.16 (.95) | 76.23 (.97)
  Physical subscale: Week 0 | 17.21 (.31) | 17.31 (.32)
  Physical subscale: Week 8: number analyzed (Participants) | 124 | 128
  Physical subscale: Week 8 | 18.96 (.33) | 18.82 (.33)
  Physical subscale: Week 20: number analyzed (Participants) | 123 | 124
  Physical subscale: Week 20 | 19.78 (.33) | 20.01 (.33)
  Physical subscale: Week 44: number analyzed (Participants) | 118 | 113
  Physical subscale: Week 44 | 19.59 (.34) | 19.55 (.35)
  Social subscale: Week 0 | 19.79 (.31) | 19.64 (.32)
  Social subscale: Week 8: number analyzed (Participants) | 124 | 128
  Social subscale: Week 8 | 19.39 (.33) | 19.69 (.33)
  Social subscale: Week 20: number analyzed (Participants) | 123 | 124
  Social subscale: Week 20 | 20.14 (.34) | 20.07 (.34)
  Social subscale: Week 44: number analyzed (Participants) | 118 | 113
  Social subscale: Week 44 | 19.76 (.34) | 19.97 (.35)
  Emotional subscale: Week 0 | 15.99 (.24) | 16.01 (.24)
  Emotional subscale: Week 8: number analyzed (Participants) | 124 | 128
  Emotional subscale: Week 8 | 17.2 (.25) | 16.75 (.25)
  Emotional subscale: Week 20: number analyzed (Participants) | 123 | 124
  Emotional subscale: Week 20 | 17.66 (.26) | 17.48 (.25)
  Emotional subscale: Week 44: number analyzed (Participants) | 118 | 113
  Emotional subscale: Week 44 | 17.6 (.26) | 17.55 (.26)
  Functional subscale: Week 0 | 16.56 (.31) | 16.59 (.31)
  Functional subscale: Week 8: number analyzed (Participants) | 124 | 128
  Functional subscale: Week 8 | 17.78 (.33) | 18.17 (.33)
  Functional subscale: Week 20: number analyzed (Participants) | 123 | 124
  Functional subscale: Week 20 | 18.58 (.33) | 19.01 (.33)
  Functional subscale: Week 44: number analyzed (Participants) | 118 | 113
  Functional subscale: Week 44 | 19.11 (.33) | 19.28 (.34)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = 0.99, Mixed Models Analysis — Overall score adjusted P = 0.99 Physical subscale adjusted P = 0.99 Social subscale adjusted P = 0.99 Emotional subscale adjusted P = 0.99 Functional subscale adjusted P = 0.99; multiple-degree-of-freedom test; Group by time interaction: Overall score: F(3,731.3)=0.03 Physical subscale: F(3,744.5)=0.23 Social subscale: F(3,740.6)=0.32 Emotional subscale: F(3,743)=0.46 Functional subscale: F(3,746.1)=0.3

6. Other Pre Specified Outcome: Coping
Description: The Brief COPE measures adaptive coping. Range for each subscale (positive reframing, active coping, planning): 2-8; higher values indicate more adaptive coping. Subscales items are summed; no total score.
Time Frame: as for outcome 4
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
score on a scale
  Active coping: Week 0 | 6.35 (.11) | 6.48 (.11)
  Active coping: Week 8: number analyzed (Participants) | 124 | 128
  Active coping: Week 8 | 6.68 (.11) | 6.58 (.11)
  Active coping: Week 20: number analyzed (Participants) | 123 | 124
  Active coping: Week 20 | 6.68 (.12) | 6.58 (.12)
  Active coping: Week 44: number analyzed (Participants) | 118 | 113
  Active coping: Week 44 | 6.55 (.12) | 6.35 (.12)
  Planning: Week 0 | 6.33 (.12) | 6.54 (.12)
  Planning: Week 8: number analyzed (Participants) | 124 | 128
  Planning: Week 8 | 6.8 (.13) | 6.58 (.12)
  Planning: Week 20: number analyzed (Participants) | 123 | 124
  Planning: Week 20 | 6.95 (.13) | 6.53 (.13)
  Planning: Week 44: number analyzed (Participants) | 118 | 113
  Planning: Week 44 | 6.52 (.13) | 6.5 (.13)
  Positive reframing: Week 0 | 6.35 (.11) | 6.48 (.11)
  Positive reframing: Week 8: number analyzed (Participants) | 124 | 128
  Positive reframing: Week 8 | 6.6 (.12) | 6.57 (.12)
  Positive reframing: Week 20: number analyzed (Participants) | 123 | 124
  Positive reframing: Week 20 | 6.58 (.12) | 6.56 (.12)
  Positive reframing: Week 44: number analyzed (Participants) | 118 | 113
  Positive reframing: Week 44 | 6.4 (.12) | 6.48 (.12)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = 0.99, Mixed Models Analysis — Active coping adjusted P = 0.99 Planning adjusted P = 0.21 Positive reframing adjusted P = 0.99; multiple-degrees-of-freedom test; Active planning: F(3,746)=0.8 Planning: F(3,744.8)=2.93 Positive reframing = F(3,742)=0.21

7. Other Pre Specified Outcome: Goal Adjustment
Description: Instrument name: Goal Disengagement and Goal Reengagement Scale (GDGRS). Range: 4 to 20 for goal disengagement and 6 to 30 for goal reengagement. Subscales: goal disengagement and goal reengagement (subscale items are averaged, no total score).
  Higher values indicate greater tendency to disengage or re-engage with goals.
Time Frame: as for outcome 4
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
score on a scale
  Disengagement: Week 0 | 10.3 (.21) | 10.6 (.22)
  Disengagement: Week 8: number analyzed (Participants) | 124 | 128
  Disengagement: Week 8 | 11.3 (.23) | 10.67 (.22)
  Disengagement: Week 20: number analyzed (Participants) | 123 | 124
  Disengagement: Week 20 | 11.29 (.23) | 10.43 (.23)
  Disengagement: Week 44: number analyzed (Participants) | 118 | 113
  Disengagement: Week 44 | 11.47 (.23) | 10.39 (.24)
  Reengagement: Week 0 | 21.26 (.27) | 21.14 (.28)
  Reengagement: Week 8: number analyzed (Participants) | 124 | 128
  Reengagement: Week 8 | 21.4 (.29) | 21.81 (.29)
  Reengagement: Week 20: number analyzed (Participants) | 123 | 124
  Reengagement: Week 20 | 22.03 (.3) | 22.01 (.29)
  Reengagement: Week 44: number analyzed (Participants) | 118 | 113
  Reengagement: Week 44 | 21.5 (.3) | 22.03 (.31)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = 0.02, Mixed Models Analysis; multiple-degrees-of-freedom test; Disengagement: F(3,741.2)=5.09 Reengagement: F(3,745.7)=0.81

8. Other Pre Specified Outcome: Distress
Description: Instrument name: Hospital Anxiety and Depression Scale (HADS). Range for each subscale (no total score): 0-21. Subscales: anxiety and depression. Higher values indicate greater anxiety and depression.
Time Frame: as for outcome 4
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 144 | 140
score on a scale
  Anxiety: Week 0 | 9.08 (.22) | 8.98 (.23)
  Anxiety: Week 8: number analyzed (Participants) | 124 | 128
  Anxiety: Week 8 | 7.79 (.24) | 7.68 (.24)
  Anxiety: Week 20: number analyzed (Participants) | 123 | 124
  Anxiety: Week 20 | 7.44 (.24) | 7.49 (.24)
  Anxiety: Week 44: number analyzed (Participants) | 118 | 113
  Anxiety: Week 44 | 7.42 (.24) | 7.19 (.25)
  Depression: Week 0 | 6.13 (.21) | 6.28 (.21)
  Depression: Week 8: number analyzed (Participants) | 124 | 128
  Depression: Week 8 | 5.17 (.22) | 5.33 (.22)
  Depression: Week 20: number analyzed (Participants) | 123 | 124
  Depression: Week 20 | 4.87 (.22) | 5.18 (.22)
  Depression: Week 44: number analyzed (Participants) | 118 | 113
  Depression: Week 44 | 5.2 (.23) | 4.89 (.23)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Other — Group by time interaction (difference in trajectory); p = 0.99, Mixed Models Analysis — Anxiety adjusted P = 0.99 Depression adjusted P = 0.99; multiple-degrees-of-freedom test; Anxiety: F(3,737.5)=0.17 Depression: F(3,733.6)=0.85

9. Other Pre Specified Outcome: Occupational Performance
Description: Instrument name: Canadian Occupational Performance Scale. The participant rates each activity with Likert scales for three characteristics: satisfaction (1- 10), performance (1-10), and importance (1 - 10).
  Interpretation: Higher values indicate higher occupational performance.
Time Frame: The overall treatment effect will be computed as the between-group difference from Session 1 (baseline) and Session 9 (approximately week 20), estimated with a linear contrast.
Population: All available data were used for the linear contrasts. See Participant Flow for reasons for missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
Number analyzed (Participants) | 139 | 136
score on a scale
  Importance: Session 1 (baseline) | 8.66 (.08) | 8.87 (.08)
  Importance: Session 9 (approximately week 20): number analyzed (Participants) | 120 | 119
  Importance: Session 9 (approximately week 20) | 8.78 (.09) | 8.75 (.09)
  Performance: Session 1 (baseline) | 4.13 (.12) | 4.29 (.12)
  Performance: Session 9 (approximately week 20): number analyzed (Participants) | 120 | 119
  Performance: Session 9 (approximately week 20) | 6.99 (.13) | 6.3 (.13)
  Satisfaction: Session 1 (baseline) | 3.74 (.14) | 3.93 (.14)
  Satisfaction: Session 9 (approximately week 20): number analyzed (Participants) | 120 | 119
  Satisfaction: Session 9 (approximately week 20) | 7.15 (.15) | 6.08 (.15)
Statistical Analysis 1: Comparison: The Behavioral Activation/ Problem Solving Intervention vs Attention Control Condition; Test type: Superiority; p = .09, Mixed Models Analysis — Importance subscale: Adjusted P = .09 Performance subscale: Adjusted P = <.001 Satisfaction subscale: Adjusted P = <.001; multiple-degrees-of-freedom test; Cohen's d = .26, 95% CI 2-sided [-.01 to 0.54] — Importance subscale: Cohen's d = 0.26 (-.01, 0.54) Performance subscale: Cohen's d = 0.60 (0.32, 0.87) Satisfaction subscale: Cohen's d = 0.76 (0.48, 1.02)

ADVERSE EVENTS:
Time Frame: 44 weeks
Arm/Group | The Behavioral Activation/ Problem Solving Intervention | Attention Control Condition
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/140
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/140
Other Adverse Events (participants affected / at risk) | 0/144 | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03915548/Prot_SAP_000.pdf